CLINICAL TRIAL: NCT03656536
Title: A Phase 3, Open-Label, Randomized, Active-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib Versus Gemcitabine Plus Cisplatin Chemotherapy in First-Line Treatment of Participants With Unresectable or Metastatic Cholangiocarcinoma With FGFR2 Rearrangement (FIGHT-302)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pemigatinib Versus Chemotherapy in Unresectable or Metastatic Cholangiocarcinoma
Acronym: FIGHT-302
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to lack of enrollment resulting from a change in the standard of care for the first-line treatment of patients with cholangiocarcinoma. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-302; 2024-513513-12-00 (Registry Identifier: EU CT Number); 2018-002894-23 (EudraCT Number)
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Unresectable Cholangiocarcinoma; Metastatic Cholangiocarcinoma
Keywords: Cholangiocarcinoma; fibroblast growth factor receptor inhibitor; FGFR; FGFR rearrangement
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pemigatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pemigatinib (Experimental)
  Interventions: Drug: Pemigatinib
- Gemcitabine + Cisplatin (Active Comparator): Participants who experience disease progression while receiving gemcitabine + cisplatin or during the follow-up period and before starting a new anticancer therapy will be eligible to cross over and receive pemigatinib.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib at the protocol-defined dose administered orally once daily as continuous therapy schedule (a cycle is 3 weeks).
  Other Names: INCB054828
  Arms: Pemigatinib
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 administered as an intravenous infusion on Days 1 and 8 of every 3-week cycle for up to 8 cycles.
  Arms: Gemcitabine + Cisplatin
Drug: Cisplatin — Cisplatin 25 mg/m^2 administered as an intravenous infusion on Days 1 and 8 of every 3-week cycle for up to 8 cycles.
  Arms: Gemcitabine + Cisplatin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pemigatinib versus gemcitabine plus cisplatin chemotherapy in first-line treatment of participants with unresectable or metastatic cholangiocarcinoma with FGFR2 rearrangement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants at least 18 years of age at the time of signing the informed consent form (ICF).
* Histologically or cytologically confirmed cholangiocarcinoma that is previously untreated and considered unresectable and/or metastatic (Stage IV per the American Joint Committee on Cancer (AJCC) Cancer Staging Manual).
* Radiographically measurable or evaluable disease by CT or MRI per RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Documented FGFR2 rearrangement.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Received prior anticancer systemic therapy for unresectable and/or metastatic disease (not including adjuvant/neo-adjuvant treatment completed at least 6 months prior to enrollment, and participants that have received treatment for locally advanced disease with trans-arterial chemoembolization or selective internal radiation therapy, if clear evidence of radiological progression is observed before enrollment, or enrolled as of Amendment 6 (or Amendment 5-JP2) and the participant received 1 cycle of gemcitabine plus cisplatin [the start of study drug {Cycle 1 Day 1} must be at least 14 days and ≤ 4 weeks {28 days} from the last dose of gemcitabine plus cisplatin]).
* Child-Pugh B and C.
* Toxicities related to prior therapy(ies) must be Common Terminology Criteria for Adverse Events (CTCAE) v5.0 ≤ Grade 1 at the time of screening.
* Concurrent anticancer therapy, other than the therapies being tested in this study.
* Participant is a candidate for potentially curative surgery.
* Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to central serous retinopathy, macular/retinal degeneration, diabetic retinopathy, retinal detachment) as confirmed by ophthalmologic examination.
* Radiation therapy administered within 4 weeks of enrollment/randomization/first dose of study treatment.
* Known central nervous system (CNS) metastases or history of uncontrolled seizures.
* Known additional malignancy that is progressing or requires active treatment (exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).
* Laboratory values at screening outside the protocol-defined range.
* History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues, such as the skin, kidney, tendons or vessels due to injury, disease, and aging, in the absence of systemic mineral imbalance).
* Significant gastrointestinal disorders that could interfere with absorption, metabolism, or excretion of pemigatinib.
* Clinically significant or uncontrolled cardiac disease.
* History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically meaningful.
* Chronic or current active infectious disease requiring systemic antibiotics or antifungal or antiviral treatment within 2 weeks prior to enrollment (participants with asymptomatic chronic infections on prophylactic treatment are allowed). Note: HIV-positive participants are allowed if all of the following criteria are met: CD4+ count ≥ 300/µL, undetectable viral load, receiving antiretroviral therapy that does not interact with study drug, and no HIV/AIDS-associated opportunistic infection in the last 12 months.
* Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study treatment. Note: Moderate CYP3A4 inhibitors are not prohibited
* Known hypersensitivity or severe reaction to pemigatinib, gemcitabine, cisplatin, or their excipients.
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 12 months
  Defined as the time from date of randomization until date of disease progression (according to Response Evaluation Criteria in Solid Tumors [RECIST] v1.1 and assessed by an independent central reviewer (ICR)) or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate | Up to approximately 12 months
  Defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by an ICR.
Overall survival | Up to approximately 12 months
  Defined as the time from date of randomization until death due to any cause.
Duration of response | Up to approximately 12 months
  Defined as the time from the date of the first assessment of CR or PR until the date of the first disease progression by an ICR per RECIST v1.1 or death, whichever occurs first.
Disease control rate | Up to approximately 12 months
  Defined as the proportion of participants who achieved best overall response of CR, PR, or stable disease (SD) per RECIST v1.1 as assessed by an ICR.
Number of treatment-emergent adverse events | Up to approximately 12 months
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Quality of Life impact as assessed by the EQ-5D-3L questionnaire | Up to 12 months
Quality of Life impact as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-30 questionnaire | Up to 12 months
Quality of Life impact as assessed by the EORTC QLQ-BIL21 questionnaire | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (215):
- United States (36):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Marin Cancer Care, Greenbrae, California
  - UC Irvine Medical Center, Orange, California
  - Georgetown University-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic-Florida, Jacksonville, Florida
  - Mount Sinai Medical Center Comprehensive Cancer Center, Miami Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Clinic Foundation Ocf Ochsner Cancer Institute Oci, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada-Twain, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - White Plains Hospital, White Plains, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Med. Ctr, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Greenville Hospital System University Medical Center Institute For Translational Oncology Research, Greenville, South Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Riverside Regional Medical Center, Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
  - Aurora Research Institute, Wauwatosa, Wisconsin
- Austria (6):
  - Landeskrankenhaus Universitatsklinikum Graz, Graz
  - Innsbruck University Hospital, Innsbruck
  - Ordensklinikum Krankenhaus Der Barmherzigen Schwestern Linz, Linz
  - Salzburger Universitatsklinikum, Salzburg
  - Landeskrankenhaus Steyr, Steyr
  - Allgemeines Krankenhaus Der Stadt Wien, Vienna
- Belgium (7):
  - Ulb Hospital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Hospital de Jolimont, Haine-st-paul
  - Az Groeninge Campus Kennedylaan, Kortrijk
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cancercare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Health Authority/Qeii Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Centre Research Institute, Montreal, Quebec
- China (20):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangdong
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou
  - Shulan Hangzhou Hospital Co Ltd, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Heilongjiang Province Cancer Hospital, Harbin
  - University of Science and Technology of China-First Affiliated Hospital (Anhui Provincial Hospital), Hefei
  - Kunming 1St People'S Hospital, Kunming
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Shandong
  - Zhongshan Hospital Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital, Shanghai
  - Sichuan Cancer Hospital, Sichuan
  - Tianjin Medical University Cancer Institute Hospital, Tianjin
  - Tongji Hospital Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Northern Jiangsu Peoples Hospital, Yangzhou
- Herlev Og Gentofte Hospital, Herlev, Denmark
- Finland (3):
  - Docrates Cancer Center, Helsinki
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (19):
  - Institut Sainte Catherine, Avignon
  - Chu Besancon Hospital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Hopital Beaujon, Clichy
  - Chu de Limoges - Hospital Dupuytren, Limoges
  - Hopital Prive Jean Mermoz, Lyon
  - Chu Hopital de La Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Antoine Laccassagne, Nice
  - Hospital Universitaire Pitie-Salpetriere, Paris
  - Hopital Europeen Georges Pompidou (Hegp), Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hospital Haut-Leveque, Pessac
  - Hospital de La Miletrie, Poitiers
  - Hopital Charles Nicolle Chu Rouen Hospital de Bois-Guillaume, Rouen
  - University Hospital of Saint Etienne, Saint-Etienne
  - Centre de Lutte Contre Le Cancer - Institut de Cancerologie de L'Ouest - Rene Gauducheau, Saint-Herblain
  - Chu Toulouse Hopital Rangueil, Toulouse
  - Chu Vandoeuvre-Les-Nancy Hopital Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (22):
  - University Medical Center Rwth Aachen, Aachen
  - Charite - Campus Virchow-Klinikum, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Universitatsklinikum Bonn Aoer, Bonn
  - Klinikum Bremen-Nord, Bremen
  - Universitatsklinikum Koln, Cologne
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Klinikum Der Johann Wolfgang Goethe University, Frankfurt am Main
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Hannover Medical School, Hanover
  - Universitaetsklinikum Des Saarlandes, Homburg / SAAR
  - Universitatsklinikum Leipzig Aor, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg
  - Otto-Von-Guericke-Universitat Magdeburg, Magdeburg
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - University Hospital Grosshadern Munich, Munich
  - Klinikum Nuernberg, Nuremberg
  - Universitaetsklinikum in Tubingen, Tübingen
  - University Hospital Tuebingen, Tübingen
  - Universitatkinikums Ulm, Ulm
- St. Vincent'S University Hospital, Dublin, Ireland
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (27):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Ospedale Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione Del Piemonte Per L'Oncologia Ircc Candiolo, Candiolo
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Ospedale Degli Infermi - Faenza, Faenza
  - Irccs Azienda Ospedaliera Universitaria San Martino, Genova
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - European Institute of Oncology, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - A.O.U. Di Modena - Policlinico, Modena
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Napoli
  - Universita Degli Studi Della Campania Luigi Vanvitelli U.O.C. Oncologia Medica, Napoli
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga Orbassano, Orbassano
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - Presidio Ospedaliero Pescara, Pescara
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
  - Istituto Nazionale Tumori Regina Elena Irccs, Roma
  - Universita Campus Bio Medico Di Roma, Rome
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
  - Centro Ricerche Cliniche Di Verona (Crc), Verona
  - San Bartolo Hospital, Vicenza
- Japan (31):
  - University of Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hyogo College of Medicine Hospital, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Teikyo University Hospital, Itabashi-ku
  - Kobe University Hospital, Kobe
  - Cancer Institute Hospital of Jfcr, Kōtoku
  - Kyoto University Hospital, Kyoto
  - Nho Shikoku Cancer Center, Matsuyama
  - Kyorin University Hospital, Mitaka-shi
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Hokkaido University Hospital, Sapporo
  - Kindai University Hospital, Sayama
  - Tohoku University Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke-shi
  - Keio University Hospital, Shinjuku-ku
  - Shizuoka Cancer Center, Shizuoka
  - Osaka University Hospital, Suita-shi
  - Toyama University Hospital, Toyama
  - Yamaguchi University Hospital, Ube
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Medical Center, Yokohama
  - Kanagawa Cancer Center, Yokohama
  - Oita University Hospital, Yufu-shi
- Netherlands (4):
  - Amsterdam University Medical Centre, Amsterdam
  - Maastricht Umc+, Maastricht
  - Erasmus Medical Center, Rotterdam
  - Umc Utrecht, Utrecht
- Oslo University Hospital, Oslo, Norway
- Spain (14):
  - Hospital Materno Teresa Herrera, A Coruña
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - HOSPITAL UNiVERSITARIO DONOSTIA, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Universitari Parc Tauli, Sabadell
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital General Universitario de Valencia, Valencia
- Karolinska Institute Universitetssjukhuset Solna, Solna, Sweden
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitatsspital Zurich, Zurich
- United Kingdom (10):
  - Aberdeen Royal Infirmary, Aberdeen
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - University Hospital Coventry and Warwickshire, Coventry
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - University College London Hospitals (Uclh), London
  - Kent Oncology Centre - Maidstone Hospital, Maidstone
  - The Christie Nhs Foundation Trust, Manchester
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Bekaii-Saab TS, Valle JW, Van Cutsem E, Rimassa L, Furuse J, Ioka T, Melisi D, Macarulla T, Bridgewater J, Wasan H, Borad MJ, Abou-Alfa GK, Jiang P, Lihou CF, Zhen H, Asatiani E, Feliz L, Vogel A. FIGHT-302: first-line pemigatinib vs gemcitabine plus cisplatin for advanced cholangiocarcinoma with FGFR2 rearrangements. Future Oncol. 2020 Oct;16(30):2385-2399. doi: 10.2217/fon-2020-0429. Epub 2020 Jul 17. PMID 32677452